CLINICAL TRIAL: NCT05345015
Title: Acute and Chronic Effects of High Frequency RF Electrical Current on Pain and Muscle Function in Individuals With Musculoskeletal Pain
Brief Title: High Frequency RF Current Effects on Muscle Pain and Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Eleftherios Kellis, Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TECAR22#1
Record Dates: First submitted 2022-04-09; First posted 2022-04-25 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Chronic Low-back Pain; Hamstring Injury; Muscle; Injury, Quadriceps (Thigh); Physical Therapy; Calf Muscle Pulled
Keywords: Sport injuries; TECAR therapy; Low back pain; Muscle injury
MeSH Terms: conditions — Wounds and Injuries; Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to an electrical energy transfer (TECAR), a Transcutaneous Electrical Stimulation (TENS) or a control (CON) group in parallel for the duration of the study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Since each group is assigned into a different intervention, masking is not possible. Outcome measures will be recorded and they will be provided codes, to ensure masking of the outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute effects (Experimental): The experimental group will receive one single session of 20-min electrical energy transfer session (Capacitive mode, 0.5 Mhz radiofrequency, intensity 40%). The TENS group will receive one 20-minute session of transcutaneous electrical stimulation (TENS, asynchronous rectangular pulse, f< 50Hz). The control (CON) group will not receive any intervention. Outcome measures will be measured prior to, immediately after, 24 and 48 hours after.
  Interventions: Device: Radiofrequency Energy Transfer; Device: Transcutaneous Nerve Stimulation
- Chronic effects (Experimental): The experimental group will receive 10 sessions of 20-min electrical energy transfer session (Capacitive mode, 0.5 Mhz radiofrequency, intensity 40%). The TENS group will receive 10 20-minute sessions of transcutaneous electrical stimulation (TENS, asynchronous rectangular pulse, f< 50Hz). The control (CON) group will not receive any intervention. Outcome measures will be measured prior to, immediately after, 3 and 6 months after.
  Interventions: Device: Radiofrequency Energy Transfer; Device: Transcutaneous Nerve Stimulation

INTERVENTIONS:
Device: Radiofrequency Energy Transfer — Radiofrequency Electrical Currents (TECAR) will be delivered using a winback system (Winback, Villeneuve-Loubet, France) propagating radiofrequency waves of 448 kHz using metallic electrodes via a coupling medium. Radiofrequencies will be used in the capacitive mode , which aims to treat superficial /soft tissues in the area. The "active" plate will be applied sequentially on the skin in the injured or painful region. The base plate will be located to the other side of the injured body region (for back thigh muscle injuries, for example, the base plate will be located on the frontal thigh area, to close the current circuit. Therapy will be applied for 20 minutes, with a target intensity of 40% and a frequency of 0.5Mhz.
  Other Names: TECAR
Device: Transcutaneous Nerve Stimulation — Transcutaneous nerve stimulation (TENS) will be delivered using a Chattanooga Intellect Advanced Combo system (Chattanooga, Hixson, TN 3 7343, USA). Two electrodes will be placed on the skin at a distance so that they cover the entire painful area. The TENS asymmetric biphasic mode (phase 300 ms, frequency 80Hz, continuous cycle) will be applied. The intensity will be adjusted between 0 and 110A, such that it is tolerable by the participant. The total application time will be 20 minutes or equal to that applied for the TECAR group.
  Other Names: TENS

SUMMARY:
The purpose of this study is to examine the acute and chronic effects of high frequency electrical current transfer (frequently called "TECAR") on pain and functional movement in individuals with a musculoskeletal injury or pain. The participants will be assigned into an experimental or a control group and outcome measures will be measured prior to, after, 24 and 48 hours following a single intervention session (Acute effects) as well as 3 and 6 months after the intervention (chronic effects).

DETAILED DESCRIPTION:
The purpose of this study is to examine the acute and chronic effects of high frequency electrical current transfer (frequently called "TECAR") on pain and functional movement in individuals with a musculoskeletal injury or pain. Participants referred for muscle strain injury (hamstring, quadriceps, gastrocnemius) or chronic low back pain will be randomly allocated into one of the three groups: an experimental group (muscle injuries), experimental group (low back pain) and a control group. The project is divided in two phases. In the first phase, the acute effects of TECAR therapy will be examined. Outcome measures will be obtained prior to, after, 24 and 48 hours following a single intervention session. The intervention consists of 20-min electrical energy transfer session (Capacitive mode, 0.5 Mhz radiofrequency, intensity 40%) or a typical transcutaneous electrical stimulation (TENS, asymmetric biphasic mode, rectangular pulse, f = 80Hz) protocol. In the chronic stage, participants will receive 10 sessions (3 times a week) receiving either protocol while outcome measurements will be obtained before, immediately, 3 and 6 months after the intervention. Analysis of variance designs will be used to compare differences in each outcome between groups at different measurement sessions. The alpha level is set to p <0.05.

ELIGIBILITY:
Muscle injury group

Inclusion Criteria:

* Acute hamstring or quadriceps or calf strain injury
* Age above 18 years

Exclusion Criteria:

* Other injury or musculoskeletal condition
* Any observed organ dysfunctions
* Receipt of medication or treatment for the past 3 months

Low back pain group

Inclusion criteria

* Pain between bottom of ribs and buttock creases
* Incidents for at least half the days in the past six months
* Visual analogue pain score equal or greater than 4/10
* Pain incidents for for less than half the days in the past six months

Exclusion Criteria:

* radiographic evidence of inflammatory disease affecting the spine
* fracture
* important genetic structure abnormality in the spine
* pregnancy
* use of medication that might influence heart rate and/or blood pressure
* psychiatric disorders
* receipt of medication or treatment for the past 3 months
* No neurologic deficits (sensory, motor, or reflexes)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain Intensity | Day before, day 0, day 1, day 2, month 3, month 6
  Visual analogue scale. Scale ranges from 0 to 10. 0 indicates no pain and 10 maximum intensity pain
Change in sit and reach test measurement | Day before, day 0, day 1, day 2, month 3, month 6
  From supine position, with the feet in contact with a wooden box and the trunk flexed, participants attempt to reach with their hands as far as posible. Score is measured in cm. A higher measurement indicates higher flexibility
Change in straight leg raising test | Day before, day 0, day 1, day 2, month 3, month 6
  From supine position, the tester raises one leg (with the knee flexed about 10-20 degrees) until discomfort is reported. The range of motion (in degrees) is stored.
Change in prone flexibility test | Day before, day 0, day 1, day 2, month 3, month 6
  From the prone position, the tester flexes the knee of the participant. The maximum range of motion is stored in degrees
Change in Oswestry index score | Day before, day 0, day 1, day 2, month 3, month 6
  A questionnaire which provides a score which reflects function in activities of daily living for those with acute or chronic back pain. It consists of 10 categories of questions, with a total sum of 50. Score is expressed as a percentage of 50, where 0% indicates no functional disability and pain. 100% indicates maximum functional disability and pain

SECONDARY OUTCOMES:
Change in single leg balance test center of pressure | Day before, day 0, day 1, day 2, month 3, month 6
  Displacement of center of pressure during a 30s single-leg standing test on a pressure platform. A greater center of pressure displacement indicates less postural stability.
Functional Assessment Scale for Acute Hamstring Injuries (FASH) | Day before, day 0, day 1, day 2, month 3, month 6
  A questionnaire for the assessment of hamstring injury severity and its impact on function of injured individuals. The questionnaire consists of 10 items, each given a score from 0 to 10, where 10 represents a high level of physical ability and 0 represents complete disability. Items scores are then added, such that a lowest total score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Eleftherios Kellis, Ph.D., Principal Investigator — Professor; Thomas Apostolou, M.D., Study Director — International Hellenic University; Paris Iakovidis, Ph.D., Principal Investigator — International Hellenic University
Locations (2):
- Greece (2):
  - Physiotherapy Clinic, Kavala
  - Laboratory of Neuromechanics, Department of Physical Education and Sport Science, Aristotle University of Thessaloniki, Serres

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paolucci T, Pezzi L, Centra AM, Giannandrea N, Bellomo RG, Saggini R. Electromagnetic Field Therapy: A Rehabilitative Perspective in the Management of Musculoskeletal Pain - A Systematic Review. J Pain Res. 2020 Jun 12;13:1385-1400. doi: 10.2147/JPR.S231778. eCollection 2020. PMID 32606905
- [Background] Paolucci T, Pezzi L, Centra MA, Porreca A, Barbato C, Bellomo RG, Saggini R. Effects of capacitive and resistive electric transfer therapy in patients with painful shoulder impingement syndrome: a comparative study. J Int Med Res. 2020 Feb;48(2):300060519883090. doi: 10.1177/0300060519883090. Epub 2019 Nov 4. PMID 31680597
- [Background] Takahashi K, Suyama T, Onodera M, Hirabayashi S, Tsuzuki N, Zhong-Shi L. Clinical Effects of Capacitive Electric Transfer Hyperthermia Therapy for Lumbago. J Phys Ther Sci. 1999;11:45-51. doi:10.1589/jpts.11.45.
- [Background] Hernandez-Bule ML, Paino CL, Trillo MA, Ubeda A. Electric stimulation at 448 kHz promotes proliferation of human mesenchymal stem cells. Cell Physiol Biochem. 2014;34(5):1741-55. doi: 10.1159/000366375. Epub 2014 Nov 12. PMID 25427571
- [Background] Kumaran B, Watson T. Thermal build-up, decay and retention responses to local therapeutic application of 448 kHz capacitive resistive monopolar radiofrequency: A prospective randomised crossover study in healthy adults. Int J Hyperthermia. 2015;31(8):883-95. doi: 10.3109/02656736.2015.1092172. Epub 2015 Nov 2. PMID 26524223
- [Background] Bretelle F, Fabre C, Golka M, Pauly V, Roth B, Bechadergue V, Blanc J. Capacitive-resistive radiofrequency therapy to treat postpartum perineal pain: A randomized study. PLoS One. 2020 Apr 27;15(4):e0231869. doi: 10.1371/journal.pone.0231869. eCollection 2020. PMID 32339169
- [Background] Fousekis K, Chrysanthopoulos G, Tsekoura M, Mandalidis D, Mylonas K, Angelopoulos P, Koumoundourou D, Billis V, Tsepis E. Posterior thigh thermal skin adaptations to radiofrequency treatment at 448 kHz applied with or without Indiba(R) fascia treatment tools. J Phys Ther Sci. 2020 Apr;32(4):292-296. doi: 10.1589/jpts.32.292. Epub 2020 Apr 2. PMID 32273653
- [Background] Tashiro Y, Hasegawa S, Yokota Y, Nishiguchi S, Fukutani N, Shirooka H, Tasaka S, Matsushita T, Matsubara K, Nakayama Y, Sonoda T, Tsuboyama T, Aoyama T. Effect of Capacitive and Resistive electric transfer on haemoglobin saturation and tissue temperature. Int J Hyperthermia. 2017 Sep;33(6):696-702. doi: 10.1080/02656736.2017.1289252. Epub 2017 Feb 19. PMID 28139939
- [Background] Yokota Y, Sonoda T, Tashiro Y, Suzuki Y, Kajiwara Y, Zeidan H, Nakayama Y, Kawagoe M, Shimoura K, Tatsumi M, Nakai K, Nishida Y, Bito T, Yoshimi S, Aoyama T. Effect of Capacitive and Resistive electric transfer on changes in muscle flexibility and lumbopelvic alignment after fatiguing exercise. J Phys Ther Sci. 2018 May;30(5):719-725. doi: 10.1589/jpts.30.719. Epub 2018 May 8. PMID 29765189
- [Background] Tashiro Y, Suzuki Y, Nakayama Y, Sonoda T, Yokota Y, Kawagoe M, Tsuboyama T, Aoyama T. The effect of Capacitive and Resistive electric transfer on non-specific chronic low back pain. Electromagn Biol Med. 2020 Oct 1;39(4):437-444. doi: 10.1080/15368378.2020.1830795. Epub 2020 Oct 6. PMID 33021115